CLINICAL TRIAL: NCT00406575
Title: A Phase II Randomized, Double Blind, Placebo-Controlled Study of Recombinant Human Relaxin in Patients With Decompensated Congestive Heart Failure
Brief Title: Recombinant Human Relaxin for the Treatment of Decompensated CHF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLX.CHF.002
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Congestive Heart Failure (CHF)
Keywords: Congestive heart failure; Relaxin; Hemodynamics; Renal function
MeSH Terms: conditions — Heart Failure | interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Participants receive diluent via continuous IV infusion for 48 hours.
  Interventions: Drug: Placebo
- Low Dose rhRlx (Experimental): Participants receive recombinant human relaxin (rhRlx) via continuous IV infusion for 48 hours at a rate of 100 µg/kg/day (corresponding to a dose of 4.2 µg/kg/hr).
  Interventions: Drug: Recombinant human relaxin (rhRlx)
- High Dose rhRlx (Experimental): Participants receive recombinant human relaxin (rhRlx) via continuous IV infusion for 48 hours at a rate of 500 µg/kg/day (corresponding to a dose of 21.0 µg/kg/hr).
  Interventions: Drug: Recombinant human relaxin (rhRlx)

INTERVENTIONS:
Drug: Placebo — Placebo was the diluent used for preparation of the 100 µg/kg/day dose of active study medication.
  Other Names: Diluent
  Arms: Placebo
Drug: Recombinant human relaxin (rhRlx) — Recombinant human relaxin (rhRlx) diluted for continuous IV infusion.
  Other Names: serelaxin; serelaxin (RLX030)
  Arms: High Dose rhRlx; Low Dose rhRlx

SUMMARY:
Two doses of relaxin will be compared to placebo for the treatment of patients with decompensated CHF

DETAILED DESCRIPTION:
Pilot clinical data suggest that recombinant human relaxin may be effective in treating patients with decompensated CHF. This study will randomize patients in blinded manner to one of two doses of intravenous relaxin or placebo. Serial evaluations will include cardiac and renal function, as well as safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization
* Decompensated chronic CHF (NYHA Class III-IV)
* LVEF < 35%
* PCWP > 22 mmHg
* CI < 2.3 L/min/m2

Exclusion Criteria:

* Acute CHF
* Acute coronary syndrome
* Hypotension or shock
* Recent stroke
* Allergy or sensitivity to test agents
* Significant confounding conditions or medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cardiac hemodynamics | Baseline through 27 hours post-infusion or discharge from the hospital.

SECONDARY OUTCOMES:
Renal function | Baseline through Day 10
  Renal function was to be assessed by evaluation of serum creatinine, creatinine clearance, BUN, uric acid, GFR, RBF, urine output, sodium clearance, and body weight.
Safety and Tolerability assessed by number of patients with adverse events (AEs) | Baseline through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dschietzig, MD, Principal Investigator — Charite Hospital, Berlin, Germany
Locations (2):
- Russia (2):
  - Russian Scientific Centre of Surgery n.a. B.V.Petrovsky of Russian Academy of Medical Sciences, Moscow
  - Educational Scientific Medical Center of the General Management Department of the President of Russian Federation. City Clinical Hospital №51, Moscow